CLINICAL TRIAL: NCT01298765
Title: A 52-Week, Open Label, Longterm Treatment Evaluation of the Safety and Efficacy of BEMA® Buprenorphine in Subjects With Moderate to Severe Chronic Pain
Brief Title: Longterm Safety Study of BEMA Buprenorphine in Subjects With Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP-305
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-03

CONDITIONS: Pain; Low Back Pain; Osteoarthritis; Neuropathic Pain
Keywords: buccal soluble film
MeSH Terms: conditions — Pain; Low Back Pain; Osteoarthritis; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEMA Buprenorphine (Experimental): buprenorphine buccal soluble film
  Interventions: Drug: BEMA Buprenorphine

INTERVENTIONS:
Drug: BEMA Buprenorphine — buccal soluble film; applied to the buccal mucosa twice daily
  Other Names: buprenorphine buccal soluble film

SUMMARY:
The purpose of this study is to determine whether BEMA Buprenorphine is safe in the treatment of chronic pain.

DETAILED DESCRIPTION:
This is an open label study of up to approximately 52 weeks duration to assess the safety and effectiveness of BEMA Buprenorphine in the management of moderate to severe chronic pain.

BEMA Buprenorphine is an oral transmucosal form of the opioid analgesic, buprenorphine hydrochloride, intended for application to the buccal mucosa. Buprenorphine is a synthetic opioid that is classified as a partial μ-receptor agonist and a Schedule III controlled substance in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-nursing female aged 18 or older
* History of moderate to severe chronic pain:

  1. Subjects completing study BUP-301 (low back pain) or
  2. Osteoarthritis or neuropathic pain, or subjects not completing study BUP-301 (low back pain), pain for ≥3 months with a pain intensity ≥5 [11 point NRS] reported at the titration period Day 0/1 visit following a washout period (opioids, NSAIDs, and muscle relaxants) of approximately 12 to 24 hours AND currently taking ≤60 mg oral morphine equivalent/day (including opioid-naïve) for 1 week or longer
* Stable health, as determined by the Investigator, on the basis of medical history, physical examination, and laboratory results so as to comply with all study procedures
* Female subjects of childbearing potential must be using a recognized effective method of birth control
* Written informed consent obtained prior to any procedure being performed

Exclusion Criteria:

* Cancer related pain
* Reflex sympathetic dystrophy or causalgia (complex regional pain syndrome), acute spinal cord compression, cauda equina compression, acute nerve root compression, meningitis, or discitis
* Surgical procedure for pain within 2 months, or nerve/plexus block within 4 weeks, prior to titration period Day 0/1 visit
* History of severe emesis with opioids
* Clinically significant sleep apnea in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Finn, PharmD, Study Director — BioDelivery Sciences International
Locations (26):
- United States (26):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Arcadia, California
  - Fresno, California
  - La Jolla, California
  - Long Beach, California
  - Westminster, Colorado
  - DeLand, Florida
  - Jupiter, Florida
  - Plantation, Florida
  - Port Orange, Florida
  - Marietta, Georgia
  - Bloomington, Illinois
  - Evansville, Indiana
  - Leawood, Kansas
  - Watertown, Massachusetts
  - Las Vegas, Nevada
  - New York, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Altoona, Pennsylvania
  - Austin, Texas
  - El Paso, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- BEMA Buproneorphine Overall: buprenorphine buccal soluble film
  BEMA Buprenorphine; buccal soluble film; applied to the buccal mucosa twice daily
Period: Titration Period
Arm/Group | BEMA Buproneorphine Overall
Started | 302
Completed | 226
Not Completed | 76
Not completed — Adverse Event | 26
Not completed — Death | 1
Not completed — Lack of Efficacy | 21
Not completed — Lost to Follow-up | 9
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 10
Not completed — Other: Not Lack of Analgesic Effect | 8
Period: Long-Term Treatment Period
Arm/Group | BEMA Buproneorphine Overall
Started | 226
Completed | 127
Not Completed | 99
Not completed — Adverse Event | 19
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 19
Not completed — Physician Decision | 1
Not completed — Other: Not Lack of Analgesic Effect | 46

BASELINE CHARACTERISTICS:
Groups:
- BEMA Buproneorphine Overall: buprenorphine buccal soluble film
  BEMA Buprenorphine (All Doses): buccal soluble film; applied to the buccal mucosa twice daily
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 235
  >=65 years | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (12.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183
  Male | 119
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 58
  White | 237
  More than one race | 0
  Unknown or Not Reported | 2
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 92.86 (22.250)
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 169.14 (10.540)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 32.226 (6.8542)
NRS Pain Score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: The NRS Pain intensity score is a segmented version of a visual analog scale used to measure pain. The scale is from 0 (no pain) to 10. Scores between greater than 0 and 3 are considered mild pain, scores from greater than 3 to 6 are moderate and greater than 6 to 10 are severe. The daily average is calculated and used as baseline.
  units on a scale | 3.3 (1.94)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in NRS Pain Intensity
Description: The NRS Pain intensity score is a segmented version of a visual analog scale used to measure pain. The scale is from 0 (no pain) to 10. Scores between greater than 0 and 3 are considered mild pain, scores from greater than 3 to 6 are moderate and greater than 6 to 10 are severe. The daily average is calculated and used to calculate the change from baseline at week 52.
Time Frame: Baseline up to approximately Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 127
units on a scale | -0.24 (1.803)

2. Secondary Outcome: Patient Global Impression of Change in Pain Intensity
Description: Patient Global Impression of Change in Pain Intensity at Week 28 as measured by a 7 point scale. Patients measure their improvement from 7='very much improved', 6='much improved', 5='minimally improved', 4='no change', 3='minimally worse', 2='much worse', 1='very much worse'.
Time Frame: Baseline to Week 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 98
units on a scale | 5.5 (1.31)

3. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication/Global Satisfaction
Description: Treatment Satisfaction Questionnaire for Medication/Global Satisfaction at Week 28. Patients complete a 14 item questionaire that measures 4 scales based on side effects, effectiveness, convenience and global satisfaction. All items have either five or seven responses (except item 4), scored from one (least satisfied) to five or seven (most satisfied). The 7-item scales have a non-neutral midpoint, such that there are more positive response options than negative response options. Item scores are summed to give four domain scores, which are in turn transformed to a scale of 0-100. Item 4 was not included for scoring. If an item score is missing and half of the items in the domain are complete, domain scores may be imputed from the person-specific mean score of completed items
Time Frame: Baseline to Week 28
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 97
units on a scale | 76.6 (15.93)

4. Secondary Outcome: Subjects Overall Satisfaction With Study Drug
Description: Subjects Overall Satisfaction with Study Drug as measured on a 5 point scale, with 1 being not satisfied and 5 being very satisified.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 122
units on a scale | 4.1 (0.80)

5. Secondary Outcome: Investigator's Overall Satisfaction With Study Drug
Description: Investigator's Overall Satisfaction with Study Drug measured on a 5-point scale, with 1 being not satisfied and 5 being very satisfied.
Time Frame: Baseline to Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BEMA Buproneorphine Overall
Number analyzed (Participants) | 122
units on a scale | 4.2 (0.78)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Adverse Events that are considered treatment-emergent that occurred during the titration period.
Arm/Group | BEMA Buproneorphine Overall
Serious Adverse Events (participants affected / at risk) | 4/302
Other Adverse Events (participants affected / at risk) | 31/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEMA Buproneorphine Overall (N=302)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BEMA Buproneorphine Overall (N=302)
Nausea (Gastrointestinal disorders) | 9 (9)
Arrhythmia (Cardiac disorders) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Irritability (General disorders) | 2 (2)
Wound Infection Staphylococcal (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Epicondylitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1)
Cognitive Disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Somnolence (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No